CLINICAL TRIAL: NCT05706220
Title: Visual Processing Speed and Objective Analysis of Supranuclear Ocular Movements Control in Multiple Sclerosis Patients and Its Relationship With OCT and Reading Difficulties
Brief Title: Visual Processing Speed and Objective Analysis of Ocular Movements in Multiple Sclerosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Collaborators: Fundación Eugenio Rodríguez Pascual (Unknown); Hospital del Rio Hortega (Other)
Responsible Party: Sponsor
Other Study IDs: 22-PI045
Record Dates: First submitted 2022-11-28; First posted 2023-01-31 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome; Relapsing Remitting Multiple Sclerosis; Progressive Multiple Sclerosis
Keywords: ocular motility disorders; eye movement; eye tracking; microperimetry; fixational eye movements; visual processing speed; optical coherence tomography
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Ocular Motility Disorders | interventions — Eye-Tracking Technology; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Control group: * Ophthalmologic examination (best-corrected visual acuity, cover and uncover tests, slit-lamp biomicroscopy, funduscopy)
  * Eye movement recording with the Tobii™ Pro Nano hardware package eye-tracking system and Tobii™ Pro Lab - full edition software
  * Visual processing speed
  * Microperimetry
  * Optical coherence tomography
  Interventions: Diagnostic Test: Eye tracking; Diagnostic Test: Microperimetry; Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Visual processing speed test
- Clinically Isolated Syndrome Patients: * Ophthalmologic examination
  * Eye movement recording with the Tobii™ Pro Nano hardware package eye-tracking system and Tobii™ Pro Lab - full edition software
  * Visual processing speed
  * Microperimetry
  * Optical coherence tomography
  * Patients with a history of optic neuritis will undergo additional tests at the discretion of the researcher (e.g. visual field, FarnsworthTest)
  Interventions: Diagnostic Test: Eye tracking; Diagnostic Test: Microperimetry; Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Visual processing speed test
- Relapsing-remitting Multiple Sclerosis Patients: * Ophthalmologic examination (best-corrected visual acuity, cover and uncover tests, slit-lamp biomicroscopy, funduscopy)
  * Eye movement recording with the Tobii™ Pro Nano hardware package eye-tracking system and Tobii™ Pro Lab - full edition software
  * Visual processing speed
  * Microperimetry
  * Optical coherence tomography
  * Patients with a history of optic neuritis will undergo additional tests at the discretion of the researcher (e.g. visual field, FarnsworthTest)
  Interventions: Diagnostic Test: Eye tracking; Diagnostic Test: Microperimetry; Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Visual processing speed test
- Primary Progressive Multiple Sclerosis Patients: * Ophthalmologic examination (best-corrected visual acuity, cover and uncover tests, slit-lamp biomicroscopy, funduscopy)
  * Eye movement recording with the Tobii™ Pro Nano hardware package eye-tracking system and Tobii™ Pro Lab - full edition software
  * Visual processing speed
  * Microperimetry
  * Patients with a history of optic neuritis will undergo additional tests at the discretion of the researcher (e.g. visual field, FarnsworthTest)
  * Optical coherence tomography
  Interventions: Diagnostic Test: Eye tracking; Diagnostic Test: Microperimetry; Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Visual processing speed test

INTERVENTIONS:
Diagnostic Test: Eye tracking — Eye tracker will be used to evaluate eye movements
  Other Names: Tobii™ Pro Nano hardware package eye-tracking system and Tobii™ Pro Lab - full edition software
Diagnostic Test: Microperimetry — Perimetric examination with Expert Exam strategy Microperimetry be used for fixation test
  Other Names: Macular Integrity Assessment (MAIA™, Centervue, Padova, Italy)
Diagnostic Test: Optical coherence tomography (OCT) — Macular Cube 512x128 or 200x200 scan. OCT will be used to analysis of retinal nerve fiber layer, ganglion cell complex and ganglion-cell/inner plexiform layer
  Other Names: Cirrus High definition (HD) - OCT 5000® ,Carl Zeiss Meditec, Dublin,California, USA
Diagnostic Test: Visual processing speed test — Visual processing speed test will be used for assessing subject visual stimulus search and reach times.
  Thirty-two different everyday visual stimuli divided in four complexity groups that were presented along 8 radial visual field positions at three different eccentricities.

SUMMARY:
This project aims to analyze ocular motility problems, visual processing speed and microperimetry, and their relationship with consolidated retinal structural biomarkers (optical coherence tomography, OCT) in patients with Multiple Sclerosis w/w reading complaints comparing with healthy subjects.

DETAILED DESCRIPTION:
Anamnesis, ophthalmological medical history including difficulties in reading with appropriate glasses.

The following protocol will be applied:

* Comprehensive eye examination
* Stereopsis
* Primary gaze position
* Cover test: far and near
* Vergence and version eye movements
* Presence of nystagmus
* Far and near best corrected visual acuity, with updated refraction

  -.Pupillary light reflex
* Biomicroscopy of the anterior pole
* Intraocular pressure
* Recording of eye movements during two standardized tests: International Reading Speed Texts test (IReST®) and Developmental Eye Movement Test (DEM™) with Tobii™ Pro Nano hardware package eye-tracking system and Tobii™ Pro Lab - full edition software.
* Visual processing speed
* Microperimetry
* Optical coherence tomography
* Eye fundus
* Patients with a history of clinical optic neuritis will additionally undergo contrast sensitivity tests, the Farnsworth® test (Farnsworth test 28 Hue x 100) and normal monocular perimetry using the standard Swedish Interactive Thresholding Algorithm (SITA-central 24-2) perimeter test. Humphrey® (Humphrey visual field analyser) and other tests at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis
* Best distant corrected visual acuity equal or greater than 0.7 (decimal scale). Glasses or soft contact lenses users.
* Best close corrected visual acuity equal to or greater than 20/30 (Snellen scale).Glasses or soft contact lenses users.

Exclusion Criteria:

* Patients with a history of acute optic neuritis (ON) and/or who experienced an episode of ON <6 months prior to the study, to avoid potential interference of papilledema with accurate peripapillary RNFL thickness measurements.
* Patients with other retinal and optic nerve diseases, advanced cataracts according to the international Lens Opacities Classification System III (LOCS III) (opacities greater than C2N2)
* Patients with other ophthalmological diseases that could affect central visual acuity
* Subjects with high refractive error (+ - 6 diopters).
* Subjects with other demyelinating disorders (neuromyelitis optica or acute disseminated encephalomyelitis).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Control group (healthy volonteers) and patients with Multiple Sclerosis
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Eye Tracking Data | 24 Hours
  Characteristics of eye movements recorded with the eye tracker system during reading tests
Values for Visual Processing Speed (VPS) | 24 Hours
  VPS will be assessing subject visual stimulus search reaction time (S-RT) and reach reaction time (R-RT), measured in seconds. Thirty-two different everyday visual stimuli were divided in four complexity groups that were presented along 8 radial visual field positions at three different eccentricities (10º, 20º y 30º)
Retinal sensitivity assessed by microperimetry | 24 Hours
  Sensitivity and fixation analysis with microperimetry
Values for OCT neuroretinal and peripapillary parameters | 24 Hours
  OCT assessment will be by spectral domain-optical coherence tomography to assess the retinal nerve fiber layer thickness and macular volume in humans

SECONDARY OUTCOMES:
Fixations recorded with the eye tracker system | 24 Hours
  number of fixations, duration in milliseconds
Saccades recorded with the eye tracker system | 24 Hours
  number of saccades, duration in milliseconds
Fixation assessment with microperimetry | 24 Hours
  Fixation assessment: P1, P2 fixation points (indexes P1 and P2)
Bivariate Contour Ellipse Area (BCEA) analysis with microperimetry | 24 Hours
  BCEA assessment: areas BCEA 63, BCEA 95
Preferred Retinal Locus (PRL) analysis with microperimetry | 24 Hours
  PRL assessment: Low-PRL, PRL High
Analysis of the macular integrity (MI) with microperimetry | 24 Hours
  MI assessment: macular integrity index
Ganglion Cell Layer measurement (GCL: Macular OCT) | 24 Hours
  Optical Coherence Tomography (OCT) will be used to assess the GCL of patients with multiple sclerosis
Retinal Nerve Fiber Layer measurement (RNFL: peri-papillary OCT) | 24 Hours
  Optical Coherence Tomography (OCT) will be used to assess the RNFL of patients with multiple sclerosis
Macular ganglion cell-inner plexiform layer thickness measurement (GCIPL) | 24 Hours
  Optical Coherence Tomography (OCT) will be used to assess the GCIPL of patients with multiple sclerosis

CONTACTS AND LOCATIONS:
Locations (1):
- IOBA - Universidad de Valladolid, Valladolid, Valladolid, Spain